CLINICAL TRIAL: NCT06834529
Title: Safety and Efficacy of CAR2219 CAR-T Cells in Treatment of Relapsed/refractory CD19/CD22 Positive B Cell Leukemia and Lymphoma
Brief Title: CAR2219 CAR-T Cells for the Treatment of R/R B Cell Leukemia and Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR2219-XYBYXB
Record Dates: First submitted 2025-01-17; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Relapsed or Refractory B Cell Leukemia and Lymphoma
Keywords: CAR-T; B cell Leukemia; B cell Lymphoma; CD19/CD22
MeSH Terms: conditions — Recurrence; Leukemia, B-Cell; Lymphoma; Lymphoma, B-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- This is a single arm treatment of CAR2219 CAR-T cell. (Experimental): Experimental: CAR2219-T cells Therapy Investigational product: CAR2219-T cells Route of administration: Intravenous injection Lymphodepleting chemotherapy regimen: A combination of fludarabine and cyclophosphamide will be administered prior to the infusion of CD2219-CAR-T cells.
  Interventions: Biological: Autologous or donor's anti-CD19 and anti-CD22 dual specific CAR-T Cells Drug: Fludarabine and Cyclophosphamide.
  Interventions: Genetic: CAR2219-T cells

INTERVENTIONS:
Genetic: CAR2219-T cells — Genetic: CAR2219-T cells Each subject will be infused with single dose of CD2219-CAR-T cells. A classic "3+3" dose escalation will be employed. The low dose is 5×10^5 /kg, the medium dose is 1×10^6 /kg, and the high dose is 2×10^6 /kg.
  Drug: Fludarabine Fludarabine will be given at a dose of 30 mg/m2/day intravenously (IV) for 3 days prior to the infusion of CD2219-CAR-T cells.
  Drug: Cyclophosphamide Cyclophosphamide will be given at a dose of 300 mg/m2/day intravenously (IV) for 3 days prior to the infusion of CD2219-CAR-T cells.
  Other Names: Fludarabine; Cyclophosphamide

SUMMARY:
This is a single arm study to evaluate the safety and efficacy of CAR2219 CAR-T cells in the treatment of relapsed/refractory CD19/CD22 positive B cell Leukemia and Lymphoma.

DETAILED DESCRIPTION:
This study is an exploratory clinical trial of a single-arm, open, single-center treatment of CAR2219 CAR-T cell. 20 subjects with relapsed or refractory CD19/ CD22 positive B-cell Leukemia and Lymphoma will be enrolled and received CAR2219 CAR T cells injection therapy, and related data such as adverse reactions and therapeutic effects after medication were followed up. To evaluate its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Relapsed/refractory CD19/CD22 positive B cell Leukemia or Lymphoma must be assured and meet one of the following conditions: (1) Confirmation for either CD19 or CD22 positivity using immunohistochemistry or flow cytometry; (2) B-cell tumors include the following three categories: ① B-cell acute lymphoblastic leukemia (B-ALL); Indolent B-cell lymphoma (CLL, FL, MZL, LPL, HCL); Aggressive B-cell lymphoma (DLBCL, BL, MCL) (3) Refractory/recurrent B-ALL (include one of the following situations) : ① relapse within 12 months after the first remission; ② The first refractory patients who did not achieve complete remission after 2 cycles of standard chemotherapy regimen; ③ Failure to achieve complete remission or relapse after first-line or multi-line salvage chemotherapy; ④ Recurrence after hematopoietic stem cell transplantation. (4) Refractory/recurrent B-cell lymphoma (meeting the requirements of 1 of the first 4 below plus 5) : ① After 4 courses of chemotherapy prescribed by the standard protocol, the tumor has shrunk by less than 50% or the disease progression(PD); ② CR reached after standard chemotherapy, but relapse occurred within 12 months; ③ Two or more recurrence after CR; ④ Recurrence after hematopoietic stem cell transplantation; ⑤Patients must have received rituximab or another anti-CD20 monoclonal antibody (unless Investigator determines that tumor is CD20-negative) and an anthracycline-containing chemotherapy regimen.
3. All genders, ages: 14 to 75 years
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2.
5. Life expectancy ≥3 months;
6. HGB≥70g/L
7. Liver,kidney function and cardiopulmonary function meet the following requirements: (1) creatinine ≤1.5×ULN; (2) left ventricular ejection fraction≥50%; (3) Oxygen saturation >90%; (4) Total bilirubin ≤1.5×ULN, ALT and AST≤2.5×ULN;
8. Participants agreed to use contraception from the time of informed consent until 1 year after CAR-T cell infusion."

Exclusion Criteria:

1. Severe heart failure with left ventricular ejection fraction <50%;
2. A history of severe lung function impairment;
3. Combined with other advanced malignant tumors;
4. Complicated with severe infection that could not be effectively controlled;
5. Severe autoimmune disease or congenital immune deficiency;
6. Active hepatitis (hepatitis B virus DNA [HBV-DNA] or hepatitis C virus RNA [HCV-RNA] test results above the lower limit of detection);
7. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), or syphilis infection;
8. History of severe allergy to biological products (including antibiotics);
9. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) patients with acute graft-versus-host reaction (GVHD) one month after immunosuppressant withdrawal;
10. Patients with other serious physical or mental illnesses or laboratory abnormalities that could increase the risk of participating in the study or interfere with the results of the study, and those who were deemed by the investigator to be unsuitable for participation in the study.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
According to the incidence of treatment-related adverse events (AEs) to evaluate the safetyof CAR2219 CAR-T cells in the treatment of relapsed/refractory CD19+CD22+ B-cell Leukemia and Lymphoma. | up to 2 years
  Incidence of treatment-related adverse events (AEs) Description: Number and severity of adverse events graded according to CTCAE v5.0, including cytokine release syndrome (CRS) graded by ASTCT criteria and immune effector cell-associated neurotoxicity syndrome (ICANS) graded by ASBMT criteria
According to the determine the Maximal Tolerable Dose(MTD) to evaluate the safetyof CAR2219 CAR-T cells in the treatment of relapsed/refractory CD19+CD22+ B-cell Leukemia and Lymphoma. | MTD will be determined based on DLTs observed during the first 28 days of study treatment.

SECONDARY OUTCOMES:
According to the objective response rate (ORR) to evaluate the efficacy of CAR2219 CAR-T cells in the treatment of relapsed/refractory CD19+CD22+ B-cell Leukemia and Lymphoma. | Within 3 months following infusion of CAR2219 CAR-T cells
  Overall response rate (ORR) Description: Proportion of participants achieving complete response (CR) or partial response (PR) according to Lugano 2014 criteria for lymphomas and NCCN guidelines for leukemias, assessed via bone marrow biopsy (for leukemia) and PET/CT imaging (for lymphoma)

OTHER OUTCOMES:
CAR-T cell expansion kinetics | Up to 12 months after CAR-T treatment
  Peak CAR-T cell levels (Cmax) and persistence duration measured by flow cytometry and qPCR in peripheral blood
CAR-T cell clonality dynamics | Up to 24 months after CAR-T treatment
  Single-cell sequencing was performed to track the clonal evolution of CAR-T cells in patients at 14 days, 1 month, 3 months, 6 months, 1 year, and 2 years post-infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- the Fifth Medical Center of Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes